CLINICAL TRIAL: NCT02323568
Title: Live After an Epithelial Ovarian Cancer: Multidisciplinary Assessment of Effects and Long-term Remission in Patients Needs.
Acronym: VIVROVAIRE 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Ligue contre le cancer, France (Other); Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VIVROVAIRE 2
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2015-09

CONDITIONS: Epithelial Ovarian Cancer
Keywords: ovarian cancer; quality of life; remission more than 3 years
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gynecological consulation (Other)
  Interventions: Other: Gynecological consultation

INTERVENTIONS:
Other: Gynecological consultation

SUMMARY:
This project is part of a large multicenter multidisciplinary program that will thoroughly explore the needs and difficulties of patients with BCR as well as those involved in their care. The results of this research program will propose recommendations for better structure and understand the follow up of these patients.

From the limited data in the literature, the long-term remission in patients with ovarian cancer reported a significant and persistent fatigue, poor QoL, disorders of sexuality as well as somatic and mental illness; consumption is also a medical records for these patients.

In this context, our team has initiated a large case-control study to assess fatigue (identified major problem in the long-term remission in patients with ovarian cancer), QoL and rehabilitation of patients in remission from an epithelial ovarian cancer (regardless of the stage of cancer at diagnosis, early or advanced) 3 years after the initial treatment, compared with women of the same age without ovarian cancer or serious chronic disease , from the general population.

Patients and controls complement standardized and validated self-administered questionnaire (part 1). This study investigated 215 patients in long remission from ovarian cancer compared to 215 women of the same age without cancer. Recruitment of patients is currently underway, in close collaboration with teams from the Group GINECO very involved in this project.

Following this step, an additional component is planned: it is to offer patients who participated in part 1, a specific gynecological consultation to assess in detail the effects of the treatments in order to better meet the needs of patients .dropoff window

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years;
* Patients who received optimal treatment (surgery, chemotherapy ...)
* Patients with epithelial ovarian cancer after first-line treatment;
* Patients without other cancer (except basal cell skin carcinoma and breast cancer in situ);
* Patients without clinical relapse, biological or radiological documented at least 3 years after the initial treatment (from the end date of first line chemotherapy);
* The interviews treatments are not recognized in the period;
* Patients may be included regardless of the stage of cancer at diagnosis (early or late)
* Patients who have signed their written consent to participate in the part 2 of the study Vivrovaire;
* Patients who participated in part 1 of Vivrovaire study.

Exclusion Criteria:

* Psychiatric pathology can disrupt the conduct of the study or to prevent the interpretation of results;
* Persons deprived of liberty;
* Major subject to a measure of legal protection or unable to consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Physical sequelae measured by the functional and biological effects | At inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY, PhD, Principal Investigator — Centre François Baclesse
Locations (18):
- France (18):
  - CHU, Besançon
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - CHU, Caen
  - Centre François Baclesse, Caen
  - Centre Hospitalier, Cholet
  - CHU Grenoble, La Tronche
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut régional du cancer, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Jean Godinot, Reims
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - GHPSO, Senlis
  - Institut de cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif